CLINICAL TRIAL: NCT05967936
Title: A Prospective Randomized Study Comparing Different Types of Local Anesthesia in Outpatient Procedural Hysteroscopy
Brief Title: Paracervical Block Versus Transcervical Block in Outpatient Procedural Hysteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-12-2023-3238
Record Dates: First submitted 2023-06-19; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-06

CONDITIONS: Myoma;Uterus; Polyp Uterus
Keywords: hysteroscopy; pain; local anesthetic; ambulatory care; bupivacaine; paracervical block; transcervical block
MeSH Terms: conditions — Myofibroma; Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Multicentric, prospective, randomized trial, single-blinded, where eligible patients will be randomized to either receive paracervical or transcervical anesthesia before outpatient surgical hysteroscopy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracervical block (Active Comparator): 10cc Bupivacaine 1% at 0.5-1 cm depth of the cervicovaginal junction at 5 and 7 o'clock positions (20cc in total).
  Interventions: Drug: Bupivacaine Injection
- Transcervical block (Experimental): 10cc Bupivacaine 1% through the endocervix using an 17-gauge epidural catheter
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — evaluation of pain by using two different types of local anesthesia
  Other Names: evaluation of pain by using two different types of local anesthesia

SUMMARY:
Hysteroscopy is a minimally invasive, diagnostic and therapeutic gynecological surgical technique and the gold standard in the study of the uterine cavity. Thanks to the decrease in the diameter of hysteroscopes and to the vaginoscopic approach, anesthesia is no longer necessary in diagnostic hysteroscopy. Nevertheless, in operative hysteroscopy, given the instrumentalization and the need of cervical dilation, the use of local anesthesia, with or without sedation, is recommended. The different alternatives described in the literature are the following:

1. Cervical/ intracervical block: injection of local anesthetic into the four quadrants of the cervix.
2. Paracervical block: injection of local anesthetic in the cervicovaginal junction at 5 and 7 o'clock positions.
3. Transcervical (uterine) anesthesia: instillation of a local anesthetic agent via catheter through the cervix and into the uterine cavity.
4. Topical cervical anesthesia: application of local anesthetic in gel or spray to the cervix.

To assess the best anesthetic pathway to decrease pain during outpatient hysteroscopy, the investigators will perform a prospective multicentric study that compare two types of local anesthesia in outpatient procedural hysteroscopy: paracervical block, that is the actual gold-standard, and transcervical instillation.

DETAILED DESCRIPTION:
To assess the best anesthetic pathway to decrease pain during outpatient hysteroscopy, the investigators will perform a multicentric prospective randomized trial, single-blinded, that compares two types of local anesthesia in outpatient procedural hysteroscopy: paracervical block, that is the actual gold-standard, and transcervical instillation.

The population studied will consist in adult women with indication of an outpatient surgical hysteroscopy (myomectomy or polypectomy). Every one of them will be invited to participate the day of their procedure. In the outpatient hysteroscopy clinic, the investigators will verify inclusion and exclusion criteria, explain the objectives of the study, collect data and obtain the patient's consent.

The sample size is 242 patients (121 in each group). The study will be performed in two different centers:

* Integrated University Health Center and Social Services of the East of the Island of Montreal
* Integrated University Health Center and social services of the South Center of the Island of Montreal

Right before each procedure the patients will be randomized through anonymous and alternized enveloppes that will be distributed in each center, to either receive paracervical or transcervical anesthesia before hysteroscopy.

Each patient will receive a pre-established dose of sedative before the procedure, according to their weight: Fentanyl 0,5 mcg/kg IV and Midazolam 0,02 mg/kg. The subsequent doses will be noted.

Under sedation, with the patient in lithotomy position, a medium size speculum will be inserted. The vagina will be disinfected with chlorhexidine and the anterior lip of the cervix will be gripped with a Pozzi forceps.

According to previous randomization, each patient will receive one of the following alternatives of local anesthesia:

* Group A: Paracervical 10cc Bupivacaine 1%, without epinephrine, at 0.5-1 cm depth of the cervicovaginal junction at 5 and 7 o'clock positions (20cc in total).
* Group B: Transcervical (uterine) 10cc Bupivacaine 1% through the endocervix using an 17-Gauge epidural catheter

During the procedure (T1), the nurse will be in charge to fill the scale (to avoid bias). The patients will be given a Visual Analogue Scale (VAS) to fill 15 minutes after the procedure (before discharge), to assess pain.

For each group the investigators will calculate the average rate of pain according to the Visual Analogue Scale during and immediately after the procedure (15 minutes). The investigators will subdivide each group into pre and postmenopausal women and into nulliparous and parous women and compare their Visual Analogue Scale as well.

Statistical analysis will be performed to compare results.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* 18 years of age or older
* Indication of outpatient surgical hysteroscopy for polypectomy and myomectomy

Exclusion Criteria:

* Women under 18 years old
* Unable to understand how to score a visual analog scale pain score
* Hysteroscopy contraindication
* Patients with medical history or current status that makes outpatient procedure usafe

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the best anesthetic pathway to decrease pain during outpatient hysteroscopy | during hysteroscopy
  comparing 10 point visual analogue scale (from 0 to 10 points) between two groups of patients recieving Bupivacaine administrated through a paracervical block versus a transcervical block
To assess the best anesthetic pathway to decrease pain during outpatient hysteroscopy | 15 minutes post hysteroscopy
  comparing 10 point visual analogue scale (from 0 to 10 points) between two groups of patients recieving Bupivacaine administrated through a paracervical block versus a transcervical block

SECONDARY OUTCOMES:
Compare the pain experience based on the visual analogue scale between pre and post-menopausal patients | during hysteroscopy
  Compare the pain experience based on the 10 point visual analogue scale (from 0 to 10 points) between pre and post-menopausal patients
Compare the pain experience based on the visual analogue scale between pre and post-menopausal patients | 15 minutes post hysteroscopy
  Compare the pain experience based on the 10 point visual analogue scale (from 0 to 10 points) between pre and post-menopausal patients
Compare the pain experience based on the visual analogue scale between nulliparous and parous patients | during hysteroscopy
  Compare the pain experience based on the 10 point visual analogue scale (from 0 to 10 points) between nulliparous and parous patients
Compare the pain experience based on the visual analogue scale between nulliparous and parous patients | 15 minutes post hysteroscopy
  Compare the pain experience based on the 10 point visual analogue scale (from 0 to 10 points) between nulliparous and parous patients
To evaluate the need for an extra intravenous sedative dose. | during hysteroscopy
  Number of patients who demand an extra dose of sedative during hysteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mélissa Roy, MD, Study Director — OB-GYN
Locations (1):
- CIUSSS de l'Est de l'Île de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Readman E, Maher PJ. Pain relief and outpatient hysteroscopy: a literature review. J Am Assoc Gynecol Laparosc. 2004 Aug;11(3):315-9. doi: 10.1016/s1074-3804(05)60042-4. PMID 15559340
- [Background] Lau WC, Tam WH, Lo WK, Yuen PM. A randomised double-blind placebo-controlled trial of transcervical intrauterine local anaesthesia in outpatient hysteroscopy. BJOG. 2000 May;107(5):610-3. doi: 10.1111/j.1471-0528.2000.tb13301.x. PMID 10826574
- [Background] De Silva PM, Mahmud A, Smith PP, Clark TJ. Analgesia for Office Hysteroscopy: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2020 Jul-Aug;27(5):1034-1047. doi: 10.1016/j.jmig.2020.01.008. Epub 2020 Jan 23. PMID 31982584
- [Background] Bettocchi S, Selvaggi L. A vaginoscopic approach to reduce the pain of office hysteroscopy. J Am Assoc Gynecol Laparosc. 1997 Feb;4(2):255-8. doi: 10.1016/s1074-3804(97)80019-9. PMID 9050737
- [Background] Cicinelli E, Didonna T, Ambrosi G, Schonauer LM, Fiore G, Matteo MG. Topical anaesthesia for diagnostic hysteroscopy and endometrial biopsy in postmenopausal women: a randomised placebo-controlled double-blind study. Br J Obstet Gynaecol. 1997 Mar;104(3):316-9. doi: 10.1111/j.1471-0528.1997.tb11460.x. PMID 9091008
- [Background] Lau WC, Lo WK, Tam WH, Yuen PM. Paracervical anaesthesia in outpatient hysteroscopy: a randomised double-blind placebo-controlled trial. Br J Obstet Gynaecol. 1999 Apr;106(4):356-9. doi: 10.1111/j.1471-0528.1999.tb08274.x. PMID 10426243
- [Background] Zupi E, Luciano AA, Valli E, Marconi D, Maneschi F, Romanini C. The use of topical anesthesia in diagnostic hysteroscopy and endometrial biopsy. Fertil Steril. 1995 Feb;63(2):414-6. PMID 7843454
- [Background] Broadbent JA, Hill NC, Molnar BG, Rolfe KJ, Magos AL. Randomized placebo controlled trial to assess the role of intracervical lignocaine in outpatient hysteroscopy. Br J Obstet Gynaecol. 1992 Sep;99(9):777-9. doi: 10.1111/j.1471-0528.1992.tb13886.x. No abstract available. PMID 1420022
- [Background] Cooper NA, Khan KS, Clark TJ. Local anaesthesia for pain control during outpatient hysteroscopy: systematic review and meta-analysis. BMJ. 2010 Mar 23;340:c1130. doi: 10.1136/bmj.c1130. PMID 20332307
- [Background] Kosus N, Kosus A, Guler A, Simavli SA, Turhan NO. Transcervical intrauterine levobupivacaine infusion or paracervical block for pain control during endometrial biopsy. Exp Ther Med. 2012 Apr;3(4):683-688. doi: 10.3892/etm.2012.463. Epub 2012 Jan 30. PMID 22969951
- [Background] Guida M, Pellicano M, Zullo F, Acunzo G, Lavitola G, Palomba S, Nappi C. Outpatient operative hysteroscopy with bipolar electrode: a prospective multicentre randomized study between local anaesthesia and conscious sedation. Hum Reprod. 2003 Apr;18(4):840-3. doi: 10.1093/humrep/deg075. PMID 12660281
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Chudnoff S, Einstein M, Levie M. Paracervical block efficacy in office hysteroscopic sterilization: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):26-34. doi: 10.1097/AOG.0b013e3181c51ace. PMID 20027030